CLINICAL TRIAL: NCT05904548
Title: Vision-MR Ablation Catheter 2.0 for Treatment of Type I Atrial Flutter
Brief Title: Atrial Flutter Ablation in the iCMR
Acronym: VISABL-AFL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imricor Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISABL-AFL
Record Dates: First submitted 2023-04-13; First posted 2023-06-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Atrial Flutter Typical
Keywords: RF Ablation; interventional Cardiac Magnetic Resonance (iCMR)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vision-MR Atrial Flutter Ablation (Experimental): Type 1 Atrial Flutter ablation performed in the iCMR with the Vision-MR Ablation Catheter 2.0 and associated Advantage-MR EP recorder and stimulator system.
  Interventions: Device: RF Ablation

INTERVENTIONS:
Device: RF Ablation — RF ablation for type I atrial flutter under iCMR guidance

SUMMARY:
The VISABL-AFL clinical investigation is a prospective, single-arm, multi-center, interventional, Investigational Device Exemption (IDE) trial. The primary objectives of VISABL-AFL are to assess the safety and efficacy of radiofrequency (RF) ablation of type-I atrial flutter performed with the Vision-MR Ablation Catheter 2.0 in the iCMR environment.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated for type I atrial flutter ablations with at least 1 documented episode of type I atrial flutter within 6 months (180 days) of enrollment
* Patient 18 years and older

Exclusion Criteria:

* Contraindications for MRI procedures
* Patients who cannot have anti-arrhythmic drugs (class I or class III) prescribed for the treatment of type I atrial flutter stopped on the day of the procedure
* Previous CTI ablation procedures
* Myocardial infarction within 60 days of enrollment
* Current unstable angina
* Cardiac surgery within 90 days of enrollment
* Any cerebral ischemic event (including transient ischemic attacks) within 6 months (180 days) of enrollment
* Thrombocytosis or thrombocytopenia
* Contraindication to anticoagulation therapy
* Currently documented intracardiac thrombus or myxoma
* Implantation of permanent leads of an implantable device in or through the right atrium within 90 days of enrollment
* Prosthetic valve through which the catheter must pass
* Interatrial baffle or patch through which the catheter must pass
* Moderate or severe tricuspid valve regurgitation or stenosis
* Uncompensated congestive heart failure
* Active systemic infection
* Pregnancy or if subject plans to become pregnant during the trial
* Uncontrolled hyperthyroidism
* Any other significant uncontrolled or unstable medical condition
* Enrollment in any concurrent study without Imricor written approval
* Life expectancy of less than or equal to 2 years (730 days) per physician opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Bi-directional block confirmation | Time of procedure, following delivery of last ablation energy delivery point
  Confirmation of bidirectional conduction block of the CTI with the Vision-MR Ablation Catheter 2.0 and Osypka HAT 500 RF generator & irrigation pump.
Primary Safety Endpoint: Composite of serious cardiovascular adverse events | 7-days post procedure
  A composite of the following serious adverse events as adjudicated by an independent clinical events committee:
  * Cardiac perforation/tamponade
  * Cerebrovascular accident (CVA)
  * Transient ischemic attack (TIA)
  * Complete heart block
  * Myocardial infarction
  * Pulmonary embolism
  * MR-related serious adverse events
  * Unanticipated device related serious adverse events
  * Death

SECONDARY OUTCOMES:
Chronic Efficacy Endpoint: Freedom from type 1 atrial flutter at 90 days | 3 months (90 days)
  The percent of subjects free of documented type I atrial flutter recurrence
Chronic Safety Endpoint: all serious adverse event rate for duration of study | 3 months (90 days)
  Rate of Serious Adverse Events during the clinical investigation as adjudicated by an independent clinical events committee

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lindborg, Study Director — Imricor Medical Systems, Inc.
Locations (6):
- United States (3):
  - Johns Hopkins University (JHU), Baltimore, Maryland
  - University of Virginia (UVA), Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- l'institut Cardiologique Paris Sud (ICPS), Massy, France
- Amsterdam University Medical Center (AUMC), Amsterdam, Netherlands
- University Hospital of Vaud (CHUV), Lausanne, Switzerland